CLINICAL TRIAL: NCT02705339
Title: Genomic Landscape of EGFR Mutant NSCLC Prior to Rociletinib and at the Time of Disease Progression Following Rociletinib
Brief Title: Rociletinib Genomic Landscape in Non-small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clovis Oncology discontinued rociletinib.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201604010
Record Dates: First submitted 2016-01-12; First posted 2016-03-10 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — rociletinib; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Rociletinib (Experimental): * Rociletinib is an oral drug which will be administered on an outpatient basis at a dose of 500 mg twice per day during each 28-day cycle.
  * After completion of cycle 1, patients who tolerate the 500 mg twice per day dose without significant adverse effect may increase dosing to 625 mg twice per day at the discretion of the investigator
  Interventions: Drug: Rociletinib; Procedure: Biopsy; Procedure: Blood draw

INTERVENTIONS:
Drug: Rociletinib
  Other Names: CO-1686
Procedure: Biopsy — Standard of care biopsies will be taken at diagnosis and at the time of disease progression
Procedure: Blood draw — -Approximately 4 teaspoons of blood will be drawn before treatment begins and at the time of disease progression to look at cell-free DNA

SUMMARY:
Though patients whose tumors harbor EGFR T790M mutation appear to benefit from rociletinib, there is a need to understand the molecular mechanisms that lead to primary and acquired resistance to rociletinib. The investigators propose to conduct a clinical trial of rociletinib of patients with EGFR-mutant NSCLC with activating EGFR mutations (including exon 19 deletion or L858R mutation), with or without EGFR T790M mutation. In these patients, pre-treatment and post-progression biopsy specimens will be subjected to genomic analysis to fully understand the clonal evolution and the molecular mechanisms underpinning treatment resistance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic stage IIIB/IV lung adenocarcinoma with known activating mutations in the EGFR TK domain (including exon 19 deletion and L858R)
* Prior EGFR TKI therapy with progression, and documented EGFR T790M mutation on tumor biopsy; however, this need not be only second line
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 2.0
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 45 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Potassium within institutional limits (supplementation allowed)
  * Magnesium within normal limits (supplementation allowed)
* Tumor tissue available and deemed adequate for genomic studies.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* Received therapeutic oral or IV antibiotics within 2 weeks prior to first day of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible.
* Symptomatic, untreated or unstable central nervous system or leptomeningeal metastases. (Patients with treated and stable brain metastases (confirmed by 2 scans at least 4 weeks apart), with no evidence of cavitation or hemorrhage in the brain lesion are eligible provided that they are asymptomatic and do not require corticosteroids.)
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to rociletinib or other agents used in the study.
* Currently receiving treatment with any medication that has the potential to prolong the QT interval and the treatment cannot be discontinued or switched to a different medication.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the previous 3 months, coronary angioplasty or stenting or bypass grafting within the past 6 months, cardiac ventricular arrhythmias requiring medication, any history of 2nd or 3rd degree atrioventricular conduction defects, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of interstitial lung disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Class II to IV heart failure as defined by the New York Heart Association functional classification system. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medial regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate, to be eligible.
* Any of the following cardiac abnormalities or history:

  * Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTcF) > 450 msec
  * Inability to measure QT interval on ECG
  * Personal or family history of long QT syndrome
  * Implantable pacemaker or implantable cardioverter defibrillator
  * Resting bradycardia < 55 beats/min
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with rociletinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Active hepatitis B virus (HBV) defined by positive hepatitis B surface antigen (HBsAg) test at screening. Patients with past or resolved HBV infection (defined by a negative HBsAg test and a positive anti-hepatitis B core antigen (anti-HBc) antibody test) are eligible. HBV DNA must be obtained in these patients prior to first day of study treatment.
* Active hepatitis C virus (HCV). Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Active tuberculosis.
* Presence of active GI disease (including GI bleeding or ulceration) or other condition that could affect GI absorption) (e.g. malabsorption syndrome, history of biliary tract disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2019-11 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Somatic genetic changes in the tumor associated with disease progression | Until the time of disease progression (estimated median of 3 months)
  -The investigators plan to conduct exome and transcriptome sequencing of tumor before therapy with rociletinib and at the time of relapse. In addition, exome sequencing of peripheral blood DNA will be done (for germ line).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Until the time of disease progression (estimated median of 3 months)
  * ORR: Percentage of patients experiencing complete response or partial response
  * Complete Response (CR): Disappearance of all target lesions and non-target lesions.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Overall survival (OS) | Until death (estimated median of 8 months)
Progression-free survival (PFS) | Until the time of progression (estimated median of 3 months)
  -PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Duration of treatment | Until the time of removal from study (estimated median of 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu